CLINICAL TRIAL: NCT01671007
Title: GLORIA - AF: Global Registry on Long-Term Oral Anti-thrombotic TReatment In PAtients With Atrial Fibrillation (Phase II/III - EU/EEA Member States)
Brief Title: GLORIA-AF Registry Program (Phase II/III - EU/EEA Member States)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.136
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this part of the Registry Program patients with non-valvular atrial fibrillation (AF) at risk for stroke are enrolled to characterize the target population and to collect real world data on important outcome events. For administrative purposes the study is divided into two protocol numbers: 1160.129 for non-EU (European Union) and non-EEA (European Economic Area) countries, and 1160.136 for EU and EEA countries. The total number of patients enrolled in both protocols is estimated to be 48,000 patients, and all these patients will be included in the data analysis for study 1160.129.

ELIGIBILITY:
Inclusion criteria:

1. Age =>18 years at enrollment
2. Male or female patient (or legally acceptable representative) willing and able to provide written informed consent
3. Patient newly diagnosed (< 3 months prior to baseline visit) with non-valvular AF and at risk for stroke.

Other inclusion criteria apply.

Exclusion criteria:

1. Presence of any mechanical heart valve, or valve disease that is expected to require valve replacement intervention;
2. Patients who have received more than 60 days of vitamin K antagonist (VKA) treatment in their lifetime;
3. AF with a generally reversible cause;
4. Patients with a medical condition other than atrial fibrillation for which chronic use of an oral anticoagulant (for example, a VKA) is indicated Other exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-valvular AF
Sampling Method: Non-Probability Sample
Enrollment: 10471 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (515):
- Austria (6):
  - Klinik Pirawarth, Therapie und Rehabilitation, Bad Pirawarth, Bad Pirawarth
  - KH der Barmherzigen Schwestern Linz, Linz
  - Kepler Univ. Klinikum Linz, Linz
  - Ordination Dr. Martin Koschutnik, Oberwart, Oberwart
  - KH d. Barmherzigen Brüder Wien, Neurologie, Vienna
  - AKH - Medical University of Vienna, Vienna
- Belgium (9):
  - Namur - HOSP St-Luc de Bouge, Bouge/Namur
  - AZ Sint-Lucas, Bruges
  - Brussels - HOSP St-Jan, Brussels
  - ULB Hopital Erasme, Brussels
  - Brussels - HOSP Europe (Ste-Elisabeth), Brussels
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Liège - HOSP CHR de la Citadelle, Liège
  - Ottignies - HOSP St-Pierre, Ottignies
  - Tienen - PRAC De Wolf, Luc, Tienen
- Bulgaria (14):
  - MHAT "Deva Maria", Dept. of Cardiology, Burgas, Burgas
  - MHAT "Dr.Stambolski", Cardiology&Intensiv Care Dept,Kazanlak, Kazanlak
  - UMHAT Sv.Georgi EAD, Plovdiv
  - MHAT, Fourth Dept. of Internal Medicine, Rousse, Rousse
  - MHAT Akta Medika OOD, Sevlievo, Sevlievo
  - Multiprofile Hospital for Active Treatment, Sliven, Sliven
  - Diagnostic & Consultancy Center "Ascendent", Sofia, Sofia
  - MHAT "National Cardiology Hosp." Cardiology Dept., Sofia, Sofia
  - University Multiprofile Hospital 'Alexandrovska', Sofia, Sofia
  - MHAT, "Vita" Surgery Department, Sofia, Sofia
  - MHAT "Tsaritsa Yoanna-ISUL" Clinic of Cardiology, Sofia, Sofia
  - UMHAT, Clinic of Cardiology, Stara Zagora, Stara Zagora
  - Medical Military Academy MHAT Varna, Varna
  - Specialized Hosp.f.Active Treatment, Cardiology Dept, Yambol, Yambol
- Croatia (9):
  - Magdalena-Special Hosp.f.Cardiovas.Surgery,Krapinske Toplice, Krapinske Toplice
  - Thalassoterapia,Rehab.of heart&lung,Cardiology Clin, Opatija, Opatija
  - Clinical Hospital Split, Split
  - General Hosp. Zadar, Clinic of Internal Med, Cardiology Dept, Zadar
  - Clinical Hosp.Merkur,Clin.Internal Med,Cardiology Dep,Zagreb, Zagreb
  - Polyclinic St. Luke, Cardiology Dept., Zagreb, Zagreb
  - Univ. Hosp. Sisters of Mercy, Cardiology Dept., Zagreb, Zagreb
  - University hospital center Zagreb, Zagreb
  - Univ. Hosp. Sisters of Mercy, Neurology Clinic, Zagreb, Zagreb
- Czechia (6):
  - Cardiology Private Practice, Brno, Brno
  - University Hospital Brno, Brno
  - Cardiocentrum, Private Practice, Kladno, Kladno
  - Cardiology Private Practice, Litovel
  - Cardiology Private Practice, Praha, Prague
  - Cardiology Private Practice, Roznov pod Radhostem, Rožnov pod Radhoštěm
- Denmark (6):
  - Forskningens Hus, Aalborg
  - Sydvestjysk Sygehus Esbjerg, Hjertemedicinsk afd., Esbjerg
  - Herlev and Gentofte Hospital, Herlev
  - Nordsjællands Hospital - Hillerød, Hillerød
  - Kolding Sygehus, Kolding
  - Odense University Hospital, Odense
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Med.Centre,Internal Med.Clin/Cardiology,Tallin, Tallinn
- France (91):
  - HOP Général, Cardio, Abbeville, Abbeville
  - HOP d'Agen, Cardio, Agen, Agen
  - HOP d'Aix en Provence, cardio, Aix-en-Provence, Aix-en-Provence
  - HOP Général, Cardio, Abbeville, Aix-en-Provence
  - HOP Louis Pasteur, Cardio, Bagnols sur Ceze, Bagnols-sur-Cèze
  - HOP Bar le Duc, Pneumo, Bar le Duc, Bar-le-Duc
  - HOP de Bayonne, Bayonne
  - HOP Jean Minjoz, Besançon
  - CAB Berdagué P, Cardio, Beziers, Béziers
  - CAB Breton Dr Nicolas, Béziers
  - HOP de Béziers, Béziers
  - CLI Tivoli, Bordeaux
  - HOP Saint-André, Bordeaux
  - HOP Ambroise Paré, Boulogne-Billancourt
  - HOP Fleyriat, GERIA, Bourg-en-Bresse, Bour-en-Bresse
  - HOP de la Cavale Blanche, Brest
  - CLI les Cedres, Cardio, Brive La Gaillarde, Brive-la-Gaillarde
  - CAB Cadinot Dr D, Broglie, Broglie
  - CAB Frappé T, MG, BRUAY LA BUISSIERE, Bruay-la-Buissière
  - HOP Saint Martin, cardio, Caen, Caen
  - HOP Côte de Nacre, Caen
  - CAB Brunschwig, Cardio, Cannes, Cannes
  - HOP William Morey, Cardio, Chalon-Sur-Saône, Chalon-sur-Saône
  - CAB Loiselet P, Cherbourg
  - HOP Gabriel-Montpied, Clermont-Ferrand
  - CAB Brunehaut M, Cardio, Clermont Ferrand, Clermont-Ferrand
  - HOP Sud Francilien, Cardio, Corbeil-Essonnes, Corbeil-Essonnes
  - HOP Sud Francilien, Corbeil-Essonnes
  - HOP Henri Mondor, Créteil
  - HOP Bocage, Dijon
  - HOP Louis Pasteur, Cardio, Dole, Dole
  - CTRE Evecquemont, Cardio, Evecquemont, Évecquemont
  - HOP du Val d'Ariège, Cardio, Foix, Foix
  - HOP Michallon, La Tronche
  - CAB Benhalima B, Cardio, Le bourget, Le Bourget
  - HOP André Mignot, Le Chesnay
  - HOP Louis Pasteur, Cardio, Le Coudray, Le Coudray
  - HOP Le Mans, Le Mans
  - CAB Phan Cao Phai, Cardio, Levallois Perret, Levallois-Perret
  - CLI Libournais, Cardio, Libourne, Libourne
  - HOP Robert Boulin, cardio, Libourne, Libourne
  - CLI de la Louviere, Lille
  - CLI le Colombier, Cardio, Limoges, Limoges
  - HOP St Joseph-St Luc, Cardio, Lyon, Lyon
  - CAB Gartenlaub O, Cardio, Maison Alfort, Maisons-Alfort
  - CAB, Salem A, Cardio, Marseille, Marseille
  - HOP Européen, Marseille
  - CAB Scala P-J, Marseille
  - CAB Scemama J, Marseille
  - CAB vial, Cardio, Marseille, Marseille
  - HOP Timone, Marseille
  - HOP des Rayettes, Martigues
  - HOP de la région d'Annecy, Cardio, Metz-Tessy, Metz-Tessy
  - CAB Dillinger J, MG, Mondelange, Mondelange
  - CLI de Montargis, Cardio, Montargis, Montargis
  - CLI du Pont de Chaume, Montauban
  - HOP Raincy Montfermeil, Cardio, Montfermeil, Montfermeil
  - HOP Arnaud de Villeneuve, Montpellier
  - CAB Prunier L, Cardio, Montreuil, Montreuil
  - HOP Central, Neuro, Nancy, Nancy
  - HOP de Courbevoie, Spécialités Med, Neuilly sur Seine, Neuilly-sur-Seine
  - CAB Jamon Y, Cardio, Nîmes, Nîmes
  - HOP Carémeau, Nîmes
  - CLI Les Franciscaines, cardio, Nïmes, Nïmes
  - HOP Orléans, Cardio, Orléans, Orléans
  - CAB Audouin P, Cardio, Paris, Paris
  - CLI Turin, Cardio, Paris, Paris
  - CAB Cohen S, Paris, Paris
  - CAB Poulain F, Paris, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Pontchaillou, Rennes
  - CAB Duvilla N, Cardio, Rouen, Rouen
  - CAB Dascotte O, Cardio, St André lez Lille, Saint-André-lez-Lille
  - CAB Lequeux B, Cardio, Saint Benoit, Saint-Benoît
  - HOP Privé de la Loire, Cardio, Saint Etienne, Saint-Etienne
  - CAB Tessier P, Cardio, St Raphael, Saint-Raphaël
  - CAB Dary P, Cardio, St-Yrieix-la-Perche, Saint-Yrieix-la-Perche
  - CAB Muller J-J, Cardio, Strasbourg, Strasbourg
  - CLI de l'Ormeau, Cardio, Tarbes, Tarbes
  - CAB Houppe Nousse MP, Cardio, Thionville, Thionville
  - HOP du Léman, Thonon-les-Bains
  - HOP Sainte Musse, Toulon
  - HOP Rangueil, Toulouse
  - HOP Cardio, Tourcoing, Tourcoing
  - CAB Leprince P, MG, Tours, Tours
  - HOP Trousseau, Tours
  - CLI Village de Santé, Cardio, Trélaze, Trélazé
  - HOP Valence, Cardio, Valence, Valence
  - HOP Bretagne Atlantique, Cardio, Vannes, Vannes
  - CAB Lejay D, MG, Vieux Condé, Vieux-Condé
  - CAB Schaupp T, MG, Vihiers, Vihiers
- Germany (76):
  - Bezirkskrankenhaus, Ansbach, Ansbach
  - Kerckhoff-Klinik, Bad Nauheim, Bad Nauheim
  - Neurologische Klinik GmbH, Bad Neustadt, Bad Neustadt/Saale
  - Sozialstiftung Bamberg, Bamberg
  - Evangelisches Elisabeth-Krankenhaus, Berlin Mitte, Berlin
  - Praxis Dr. Rieker, Berlin, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Praxis Dr. Altmann, Berlin, Berlin
  - Praxisgemeinschaft Dres. Weinrich, Berlin
  - Praxis Dr. Claus, 10969 Berlin, Berlin
  - Kardiologische Praxis Dr. Jochen Bott, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - Gesundheit Nord gGmbH | Klinikverbund Bremen, Bremen
  - Klinikum Bremerhaven, Bremerhaven
  - Herz- und Gefaesszentrum am Neumarkt, Celle
  - Gemeinschaftspraxis Dr. med. J. Sek, Chemnitz, Chemnitz
  - Klinikum Coburg gGmbH, Coburg
  - Praxis für Kardiologie, Köln, Cologne
  - HELIOS Amper Kliniken, Dachau, Dachau
  - Kardiologische Praxisgemeinschaft,Darmstadt, Darmstadt
  - Praxis Dr. Rybak, Dessau, Dessau
  - Klinikum Lippe-Detmold GmbH, Detmold
  - Kardiologischen Gemeinschaftspraxis Dinslaken, Dinslaken
  - Praxis Dr. med. Bernhard-Paul Lodde, Dortmund
  - Praxisklinik Herz und Gefäße, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Praxis für Herz-Kreislauf-Erkrankungen Zeulenroda-Greiz, Greiz
  - Asklepios Klinik St. Geort, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Harburg, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Praxis Herz im Zentrum Laske, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Ingolstadt GmbH, Ingolstadt
  - Praxis Dr. Mibach, Itzehoe, Itzehoe
  - Universitätsklinikum Jena, Jena
  - Kardiologische Gemeinschaftspraxis Kassel, Kassel
  - Praxis Dr. med. Frickel Siegfried, Kempen
  - Praxis Dr. med. Matthias Gabelmann, Kirchzarten
  - St. Antonius-Hospital, Kleve, Kleve
  - Universitätsklinikum Leipzig, Leipzig
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum Leverkusen gGmbH, Leverkusen, Leverkusen
  - Cardio Centrum Ludwigsburg, Ludwigsburg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Gemeinsachftspraxis Regner/Schmitt/Kros, Mainz, Mainz
  - Praxis Dr.med. Jens Taggeselle, Markkleeberg, Markkleeberg
  - Klinikum Memmingen, Memmingen
  - Johannes Wesling Klinikum, Minden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Praxis Dr. med. Norbert Schön, Mühldorf, Mühldorf
  - Herzzentrum ALTER HOF München, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Praxis Dr. med. Joachim Gmehling, Nuremberg
  - Klinikum Osnabrück GmbH, Osnabrück
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis Papenburg, Papenburg
  - Kardiologisches Zentrum Peine, Peine
  - Städt. Krankenhaus, Pforzheim, Pforzheim
  - Kardiologische Gemeinschaftspraxis Potsdam, Potsdam
  - Kardiologische Gemeinschaftspraxis Rostock, Rostock
  - Kreisklinikum Siegen GmbH, Siegen
  - Berufsausübungsgemeinschaft Klein /Kratochvil, Stuttgart
  - Herzklinik Ulm Gemeinschaftspraxis, Ulm
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Kardiologische Praxis, Wermsdorf, Wermsdorf
  - MedKonsil, Wiesbaden, Wiesbaden
  - Kardiologische Gemeinschaftspraxis Wittenberg, Wittenberg
  - Universitätsklinikum Würzburg, Würzburg
- Greece (18):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Euroclinic of Athens, Athens
  - "Korgialeneio-Benakeio" Hellenic Red Cross Hospital, Athens
  - Sotiria Hosp.,Hypertension Unit,3rd Clinic of Internal Med., Athens
  - Asclepion Voulas Hospital, Cardiological Clinic, Athens
  - General Hospital of Chalkida, Chalcis
  - General Hospital of Chania, Chania
  - General Hospital of Edessa, Cardiology Clinic, Edessa
  - Gen. Hosp. of Elefsina "Thriassio", Elefsina
  - University General Hospital of Heraklion, Herakleion, Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General Hospital Komotinis, Komotini
  - General University Hospital of Larissa, Larissa
  - University of Patras Medical School, Pátrai
  - General Hospital of Rhodes, Rhodes
  - Gen. Hosp. of Thessaloniki "Hippokation", Cardiology Clinic, Thessaloniki
  - "Papageorgiou" General Hospital of Thessaloniki, B' Cardiolo, Thessaloniki
  - General Panarkadiko Hospital of Tripolis, Cardiology Clinic, Tripoli
- Ireland (5):
  - Portiuncula Hospital, Ballinasloe
  - Adelaide & Meath Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
  - The Redhouse Family Practice, Mallow
- Italy (72):
  - Ospedale Riuniti Albano Genzano, Albano Laziale
  - Az. Osp. S.M. di Misericordia, Albenga
  - Az. Ospedaliere Umberto I di Ancona, Ancona
  - Ospedale Reg Umberto Parini, Aosta
  - Ospedale C. G. Mazzoni, Ascoli Piceno
  - AZ. Osp. Assisi U.O., Assisi
  - Osp. SS Filippo Nicola, Avezzano
  - Policlinico di Bari, Bari
  - Policlinico Universitario di Bari, Bari
  - Policlinico S. Orsola Malpighi, Bologna
  - A. O. G. Brotzu, Cagliari
  - Presidio Ospedaliero di Castrovillari, Castrovillari (CS)
  - P. O. "Garibaldi" - Nesima, Catania
  - A.O. Univ. Vittorio Ferrarotto S. Bambino, Catania
  - Policlinico Universitario Mater Domini, Universita di Catanzaro, Catanzaro
  - Osp. Clin. SS. Anunziata, Chieti
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona (FE)
  - Osp.S.Salvatore, Coppitto (AQ)
  - AZ. Osped. Ospedale Maggiore di Crema, Crema (CR)
  - A. Istituti Osp. di Cremona, Cremona
  - Ospedale S. Biagio, Domodossola (VB)
  - P. O. S. Maria Nuova, Florence
  - Azienda Ospedaliera Careggi, Florence
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Ospedale S. Cuore di Gesù, Gallipoli
  - Policlinico San Martino, Genova
  - Ospedale della Misericordia, Grosseto
  - Ospedale F. Veneziale, Isernia
  - Azienda Ospedaliera C. Poma, Mantova
  - Osp. Pediatrico Aprano Pasquinucci, Massa
  - Az Osp. Amico " Gaetano Fucito", Mercato San Severino (SA)
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Nuovo Ospedale Civile S. Agostino-Estense, Modena
  - Osp.Riun.Valdichiana Senese, Montepulciano Senese (SI)
  - A.O. San Gerardo di Monza, Monza (MB)
  - Ospedale Nuovo Pellegrini, Napoli
  - Ospedale Cardarelli, Napoli
  - Osp.Sacro Cuore-Don Calabria, Negrar (VR)
  - Az. Osp. San Giacomo, Novi Ligure
  - Az. Osp. San Francesco, Nuoro
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - A.O. Univ. Policlinico Giaccone, Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
  - Ospedale San Salvatore, Pesaro
  - Osp. Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - Ospedale Santa Corona Azienda Sanitaria Locale n.2 Savonese, Pietra Ligure
  - Ospedale di Cisanello, Pisa
  - Ospedale S.Tommaso dei Battuti, Portogruaro (VE)
  - P.O.S. Maria Grazie, Pozzuoli
  - Azienda Unità Sanitaria Locale di Reggio Emilia, Reggio Emilia
  - Ospedale "Giambattista Grassi, Roma
  - Pol. Universitario Tor Vergata, Roma
  - Azienda Complessa Ospedaliera Ospedale San Fiippo Neri, Roma
  - Ospedale "S. Eugenio", Roma
  - A.O. San Camillo Forlanini, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Policlinico Gemelli, Roma
  - Policlinico Casilino U.O. Cardiologia, Roma
  - Az. Osp.Madre Giuseppina Vannini-, Roma
  - Az. Osp. S.Giovanni-Addolorata, Roma
  - Ospedale S. Spirito, Roma
  - Nuovo Ospedale Civile di Sassuolo, Sassuolo
  - IRCCS Gruppo Multimedica, Sesto S.Giovanni (MI)
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - AO Città della Salute e della, Torino
  - Ospedale Mauriziano di Torino, Torino
  - Ospedale S. Maria di Ca' Foncello Azienda ULSS9 TREVISO, Treviso
  - A. O. S. Maria della Misericordia, Udine
  - A. O. Ospedale Circolo Fond. Macchi, Varese
  - Ospedale San Bortolo, Vicenza
- Latvia (3):
  - Liepaja Regional Hospital, Therapy Department, Liepāja
  - P.Stradins Clin.Univ.Hosp,Cardio.Diagnos&Outpatient Dep,Riga, Riga
  - Riga East University Hospital, Riga
- Netherlands (21):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Rijnstate Hospital, Arnhem
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Groep, Delft
  - Noordwest Ziekenhuisgroep, Den Helder
  - Deventer Ziekenhuis, Deventer
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medisch Centrum, Heerlen
  - TREANT zorggroep, Hoogeveen
  - Westfries Gasthuis, Hoorn
  - METC Academisch Ziekenhuis Maastricht/Universiteit van Maastricht, Maastricht
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Havenziekenhuis, Rotterdam
  - Zuyderland Medisch Centrum, Sittard - Geleen
  - Antonius Ziekenhuis, Sneek
  - Ziekenhuis Rivierenland, Tiel
  - VieCuri Medisch Centrum, locatie Venray, Venray
  - Isala Zwolle, Zwolle
- Norway (8):
  - Legegruppen Arendal, Arendal
  - Vestre Viken HF, Bærum sykehus, Drammen
  - Medisinsk Senter Fornebu DA, Fornebu
  - Vestre Viken, Ringerike Sykehus HF, Hønefoss
  - Sykehuset Innlandet HF, Kongsvinger, Kongsvinger
  - Sykehuset Innlandet HF, Avd. Lillehammer, Lillehammer
  - Volvat Medisinske senter, Oslo, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (14):
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - Private Practice Jacek Kowalczyk, Bytom, Bytom
  - Specialist Out-patient Clinics 'Na Gornej',Cieszyn, Cieszyn
  - Specialistic Cardiology&Hypertension Out-patient Clin,Kielce, Kielce
  - Private Practice of Heart Diseases Malgorzata Lelonek,Lodz, Lodz
  - Allmedica Sp. z.o.o, prac. Nowy Targ, Nowy Targ
  - Private Specialistic Practices, Nysa, Nysa
  - Reg.Hosp, Intern.Med.Ward w/ Intensive Cardiol.Care, Opoczno, Opoczno
  - Szpital Specjalistyczny w Pulawach, Puławy
  - Cardiology Out-patient Clinic "Cardio-Plus", Radlin, Radlin
  - Internal Medicine,Cardiol.practiceWanda&Jerzy Sudnik,Sokolka, Sokółka
  - Individual Specialist.Private Practice Dr.W.Krysiak,Szczecin, Szczecin
  - Individual Specialistic Private Practice,Dr.A.Tomasik,Zabrze, Zabrze
  - Slaskie Center Heart Disease SUM,Cardiol.&Electr.Clin.Zabrze, Zabrze
- Portugal (10):
  - Hospital Garcia de Orta, EPE, Almada
  - CHLO, EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar da Cova da Beira Hospital Pêro da Covilhã, Covilha
  - Hospital do Espírito Santo, EPE, Evora
  - Centro Hospitalar Algarve, EPE, Faro
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - CHLO, EPE - Hospital S. Francisco Xavier, Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
  - Hospital de Santiago, Setúbal
- Romania (12):
  - CMI Dr. Bogdan Minescu, Braila, Brăila
  - Emergency University Hospital, Bucharest, Bucharest
  - ILRO Medical SRL, Bucharest, Bucharest
  - Med.Centre Diagnosis,Treatm&Prev Med.Cardiol.Dept, Bucharest, Bucharest
  - SC Titan Medical SRL, Bucharest, Bucharest
  - Humanitas Medical Center, Bucharest, Bucharest
  - SC Cardiomed SRL, Cluj Napoca, Cluj-Napoca
  - SC Cardiomed SRL, Constanta, Constanța
  - S.C Cardiomed S.R.L, Craiova
  - SC Cardiomed SRL, Iasi, Iași
  - Galenus Medical Center, Targu Mures, Târgu Mureş
  - Medicorclinics, Timisoara, Timișoara
- Slovenia (2):
  - General Hospital Celje, Celje
  - Univ. Medical Centre Ljubljana, Dept. of Vascular Diseases, Ljubljana
- Spain (43):
  - Hospital A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - CAP Passeig de Maragall, Barcelona
  - Consultorio Cañaveral, Cañaveral (Cáceres)
  - Hospital Santa Lucía, Cartagena (Murcia)
  - Hospital La Princesa, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de la Arrixaca, El Palmar - Murcia
  - Hospital Universitario San Cecilio, Granada
  - Hospital Jerez de la Frontera, Jerez de La Frontera - Cádiz
  - Hospital de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Severo Ochoa, Leganes - Madrid
  - Hospital de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón y Cajal, Madrid
  - Centro de Salud Jazmin, Madrid
  - Centro de Salud Isla de Oza, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Regional Universitario de Málaga, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Costa del Sol, Marbella . Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital General Universitario de Alicante, Sant Joan d'Alacant
  - Hospital Moises Broggi, Sant Joan Despí
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital San Juan de Dios, Seville
  - Hospital Virgen del Rocío, Seville
  - ABP Salud Sevilla, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - CS Ingeniero Joaquin Benlloch, Valencia
  - Hospital Univ La Fe, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Comarcal Axarquía, Vélez-Málaga
  - Hospital Meixoeiro, Vigo
  - Hospital Povisa, Vigo
- Sweden (7):
  - Falu lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Skånes universitetssjukhus, Malmö, Malmo
  - Stockholm Heart Center AB, Stockholm
  - Danderyds Sjukhus, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Centrallasarettet, Västerås, Västerås
- United Kingdom (81):
  - Gale Farm Surgery, Acomb
  - William Harvey Hospital, Ashford
  - Axbridge and Wedmore Medical Practice, Axbridge
  - Basildon University Hospital, Basildon
  - North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath
  - Beehive Surgery, Bath
  - Birmingham City Hospital, Birmingham
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Bradgate Surgery, Bristol
  - Bristol Royal Infirmary, Bristol
  - Clevedon Riverside Group, Bristol
  - Burbage Surgery, Burbage, Hinkley
  - West Suffolk Hospital, Bury St Edmunds
  - Cumberland Infirmary, Carlisle
  - Countess of Chester Hospital, Chester
  - Castle Hill Hopsital, Cottingham
  - Pound Hill Medical Group, Crawley
  - Dorset County Hospital, Dorchester
  - Russells Hall Hospital, Dudley
  - Ninewells Hospital & Medical School, Dundee
  - University Hospital of North Durham, Durham
  - Royal Devon and Exeter Hospital, Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - The County Hospital, Hereford
  - Wycombe General Hospital, High Wycombe
  - Honiton Surgery Group - Seamark, Honiton
  - Hedon Group Practice, Hull
  - Airedale General Hospital, Keighley
  - Westmorland General Hospital, Kendal
  - Leeds General Infirmary, Leeds
  - Research Unit, Liverpool Heart and Chest Hospital, Liverpool
  - Aintree University Hospital, Liverpool
  - University Hospital Lewisham, London
  - St George's Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Luton and Dunstable University Hospital, Luton
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - St Chad's Surgery, Midsomer Norton
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital, Norwich
  - George Eliot Hospital, Nuneaton
  - Royal Oldham Hospital, Oldham
  - Perth Royal Infirmary, Perth
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Poole Hospital, Poole
  - Craigavon Area Hospital, Portadown, County Atrim
  - Royal Preston Hospital, Preston
  - Royal Berkshire Hospital, Reading
  - Alexandra Hospital, Redditch
  - Sherbourne Medical Centre, Royal Leamington Spa
  - Cape Cornwall Surgery, Saint Just, Penzance
  - The Conquest Hospital, Saint Leonards-on-Sea
  - Salisbury District Hospital, Salisbury
  - Royal Shrewsbury Hospital, Shrewsbury
  - Wexham Park Hospital, Slough
  - County Hospital, Stafford
  - Branch End Surgery, Stocksfield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay
  - South Tyneside District Hospital, Tyne-and-Wear
  - Hillingdon Hospital, Uxbridge
  - Wansford Surgery, Wansford, Peterborough
  - The Avenue Surgery, Warminster
  - Warwick Hospital, Warwick
  - Queen Elizabeth II Hospital, Welwyn Garden City
  - Westbury Group Practice, Westbury
  - Southend General Hospital, Westcliffe-on-Sea
  - Whitby Group Practice, Whitby
  - New Cross Hospital, Wolverhampton
  - Jorvik Medical Practice, York
  - York Medical Group, York
  - The York Hospital, York
  - MyHealth, Strensall Health Care Centre, York

REFERENCES:
- [Derived] Joddrell M, El-Bouri W, Harrison SL, Huisman MV, Lip GYH, Zheng Y; GLORIA-AFinvestigators. Machine learning for outcome prediction in patients with non-valvular atrial fibrillation from the GLORIA-AF registry. Sci Rep. 2024 Nov 7;14(1):27088. doi: 10.1038/s41598-024-78120-z. PMID 39511367
- [Derived] Romiti GF, Corica B, Proietti M, Mei DA, Frydenlund J, Bisson A, Boriani G, Olshansky B, Chan YH, Huisman MV, Chao TF, Lip GYH; GLORIA-AF Investigators. Patterns of oral anticoagulant use and outcomes in Asian patients with atrial fibrillation: a post-hoc analysis from the GLORIA-AF Registry. EClinicalMedicine. 2023 Aug 25;63:102039. doi: 10.1016/j.eclinm.2023.102039. eCollection 2023 Sep. PMID 37753446
- [Derived] Ding WY, Fawzy AM, Romiti GF, Proietti M, Pastori D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Validating the predictive ability of the 2MACE score for major adverse cardiovascular events in patients with atrial fibrillation: results from phase II/III of the GLORIA-AF registry. J Thromb Thrombolysis. 2024 Jan;57(1):39-49. doi: 10.1007/s11239-023-02866-y. Epub 2023 Aug 11. PMID 37566295
- [Derived] Ding WY, Lane DA, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Incidence and Risk Factors for Residual Adverse Events Despite Anticoagulation in Atrial Fibrillation: Results From Phase II/III of the GLORIA-AF Registry. J Am Heart Assoc. 2022 Aug 2;11(15):e026410. doi: 10.1161/JAHA.122.026410. Epub 2022 Jul 25. PMID 35876418
- [Derived] Ding WY, Calvert P, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Impact of early ablation of atrial fibrillation on long-term outcomes: results from phase II/III of the GLORIA-AF registry. Clin Res Cardiol. 2022 Sep;111(9):1057-1068. doi: 10.1007/s00392-022-02022-1. Epub 2022 Apr 29. PMID 35488127
- [Derived] Lip GYH, Kotalczyk A, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Marler S, Gurusamy VK, Huisman MV; GLORIA-AF Investigators. Comparative effectiveness and safety of non-vitamin K antagonists for atrial fibrillation in clinical practice: GLORIA-AF Registry. Clin Res Cardiol. 2022 May;111(5):560-573. doi: 10.1007/s00392-022-01996-2. Epub 2022 Mar 16. PMID 35294625
- [Derived] Huisman MV, Teutsch C, Lu S, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Lohmann R, Gurusamy VK, Bartels DB, Lip GYH; GLORIA-AF Investigators. Dabigatran versus vitamin K antagonists for atrial fibrillation in clinical practice: final outcomes from Phase III of the GLORIA-AF registry. Clin Res Cardiol. 2022 May;111(5):548-559. doi: 10.1007/s00392-021-01957-1. Epub 2022 Mar 16. PMID 35294623
- [Derived] Bayer V, Kotalczyk A, Kea B, Teutsch C, Larsen P, Button D, Huisman MV, Lip GYH, Olshansky B. Global Oral Anticoagulation Use Varies by Region in Patients With Recent Diagnosis of Atrial Fibrillation: The GLORIA-AF Phase III Registry. J Am Heart Assoc. 2022 Mar 15;11(6):e023907. doi: 10.1161/JAHA.121.023907. Epub 2022 Mar 4. PMID 35243870
- [Derived] Ntaios G, Huisman MV, Diener HC, Halperin JL, Teutsch C, Marler S, Gurusamy VK, Thompson M, Lip GYH, Olshansky B; GLORIA-AF Investigators. Anticoagulant selection in relation to the SAMe-TT2R2 score in patients with atrial fibrillation: The GLORIA-AF registry. Hellenic J Cardiol. 2021 Mar-Apr;62(2):152-157. doi: 10.1016/j.hjc.2020.11.009. Epub 2020 Dec 15. PMID 33338644
- [Derived] Huisman MV, Rothman KJ, Paquette M, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Zint K, Elsaesser A, Lu S, Bartels DB, Lip GYH; GLORIA-AF Investigators. Two-year follow-up of patients treated with dabigatran for stroke prevention in atrial fibrillation: Global Registry on Long-Term Antithrombotic Treatment in Patients with Atrial Fibrillation (GLORIA-AF) registry. Am Heart J. 2018 Apr;198:55-63. doi: 10.1016/j.ahj.2017.08.018. Epub 2017 Aug 31. PMID 29653649
- [Derived] Huisman MV, Lip GY, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Teutsch C, Zint K, Ackermann D, Clemens A, Bartels DB. Design and rationale of Global Registry on Long-Term Oral Antithrombotic Treatment in Patients with Atrial Fibrillation: a global registry program on long-term oral antithrombotic treatment in patients with atrial fibrillation. Am Heart J. 2014 Mar;167(3):329-34. doi: 10.1016/j.ahj.2013.12.006. Epub 2013 Dec 19. PMID 24576516
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated characteristics of patients with non-valvular atrial fibrillation influencing the choice of antithrombotic treatment for the prevention of stroke, and the safety and effectiveness of dabigatran versus Vitamin K Antagonist for up to 3-year follow-up period.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the study. Subjects attended a participating site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Dabigatran Etexilate - Baseline: Patients who were prescribed Dabigatran etexilate at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Vitamin K Antagonist (VKA) - Baseline: Patients who were prescribed Vitamin K Antagonist (VKA) at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Rivaroxaban - Baseline: Patients who were prescribed Rivaroxaban at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Apixaban - Baseline: Patients who were prescribed Apixaban at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Edoxaban - Baseline: Patients who were prescribed Edoxaban at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Acetylsalicylic Acid (ASA) - Baseline: Patients who were prescribed Acetylsalicylic acid (ASA) at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Antiplts Other Than ASA - Baseline: Patients who were prescribed Antiplts other than Acetylsalicylic acid (ASA) at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- No Treatment - Baseline: Patients who were prescribed no treatment at baseline were included in this group. Patients can take other Antithrombotic treatments later during the study.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
- Combinations With Oral Anticoagulants - Baseline: Patients who were prescribed the treatments with combinations with oral anticoagulants at baseline were included in this group. This group of patients were not included in the safety analysis as no specific treatment can be defined.
  Patients who were newly diagnosed non-valvular Atrial Fibrillation (AF) less than 3 months before the baseline visits (less than 4.5 months before baseline visit for Latin America) and who were at risk for stroke in a real-life setting. Antithrombotic treatments were used according to local practice for stroke prevention. The choice of antithrombotic agent and dosing was at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline | Rivaroxaban - Baseline | Apixaban - Baseline | Edoxaban - Baseline | Acetylsalicylic Acid (ASA) - Baseline | Antiplts Other Than ASA - Baseline | No Treatment - Baseline | Combinations With Oral Anticoagulants - Baseline
Started | 2089 | 2834 | 2033 | 2214 | 180 | 513 | 80 | 526 | 2
All Eligible | 2066 | 2758 | 2008 | 2197 | 180 | 507 | 79 | 507 | 2
Completed | 1768 | 2183 | 1667 | 1846 | 155 | 401 | 59 | 394 | 2
Not Completed | 321 | 651 | 366 | 368 | 25 | 112 | 21 | 132 | 0
Not completed — Other reasons than listed | 166 | 373 | 197 | 228 | 14 | 71 | 17 | 66 | 0
Not completed — Withdrawal by Subject | 36 | 59 | 53 | 58 | 4 | 15 | 1 | 19 | 0
Not completed — Lost to Follow-up | 93 | 142 | 91 | 63 | 7 | 20 | 2 | 28 | 0
Not completed — No end of study case report form | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Not eligible | 23 | 76 | 25 | 17 | 0 | 6 | 1 | 19 | 0

BASELINE CHARACTERISTICS:
Population: All eligible: All patients who were enrolled and eligible (i.e. did not have any important. protocol violation(s) and who met certain data cleaning requirements).
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline | Rivaroxaban - Baseline | Apixaban - Baseline | Edoxaban - Baseline | Acetylsalicylic Acid (ASA) - Baseline | Antiplts Other Than ASA - Baseline | No Treatment - Baseline | Combinations With Oral Anticoagulants - Baseline | Total
Number analyzed (Participants) | 2066 | 2758 | 2008 | 2197 | 180 | 507 | 79 | 507 | 2 | 10304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.3 (9.4) | 72.8 (9.5) | 71.1 (10.1) | 73.3 (9.8) | 73.3 (9.2) | 70.5 (12.4) | 74.2 (11.1) | 68.7 (12.5) | 71.5 (0.7) | 72.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 942 | 1252 | 894 | 990 | 86 | 234 | 25 | 246 | 1 | 4670
  Male | 1124 | 1506 | 1114 | 1207 | 94 | 273 | 54 | 261 | 1 | 5634
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 14 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 21
  Asian | 4 | 4 | 7 | 7 | 0 | 2 | 0 | 1 | 0 | 25
  Black/African American | 4 | 6 | 9 | 9 | 1 | 1 | 1 | 0 | 0 | 31
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1792 | 2526 | 1735 | 1835 | 178 | 430 | 75 | 482 | 2 | 9055
  Other | 7 | 9 | 4 | 6 | 1 | 2 | 0 | 2 | 0 | 31
  Missing | 254 | 199 | 253 | 339 | 0 | 71 | 3 | 22 | 0 | 1141

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction, Life-threatening Bleeding Events and Vascular Death)
Description: Incidence rate of composite outcome which includes events of Stroke, systemic embolism, myocardial infarction, life-threatening bleeding events and vascular death on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only. In case of multiple events for a patient, the first event was considered. Unknown death was imputed by multiple imputation. The average of the 20 incidence rates from the 20 imputed datasets were used to obtain the point estimate of the incidence rate that is reported here. The bootstrapping approach was used to obtain the 95% confidence interval of the incidence rate.
Time Frame: From baseline visit until end of initial treatment regimen episode (minimum date of permanent stop of DE + 3 days/ VKA+ 6 days, start date of other treatments - 1 day, and date of study completion/discontinuation), up to 3 years.
Population: Restricted patient set: the set consists of all eligible patients who were within the region of propensity score (PS) overlap excluding patients in the non-overlapping tails of the propensity score distribution. The restricted patient set was defined for dabigatran etexilate and vitamin K antagonist patients only.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 2.30 [1.86 to 2.73] | 3.02 [2.54 to 3.54]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous stroke/transient ischaemic attack/systemic embolism, previous myocardial infarction, abnormal kidney function and concomitant antiplatelets use; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.64 to 1.08] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

2. Primary Outcome: Incidence Rate of Vascular Composite Outcome (Stroke, Systemic Embolism, Myocardial Infarction and Vascular Death)
Description: Incidence rate of vascular composite outcome including events of stroke, systemic embolism, myocardial infarction and vascular death on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only. In case of multiple events for a patient, the first event was considered. Unknown death was imputed by multiple imputation. The average of the 20 incidence rates from the 20 imputed datasets were used to obtain the point estimate of the incidence rate that is reported here. The bootstrapping approach was used to obtain the 95% confidence interval of the incidence rate.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 1.91 [1.52 to 2.32] | 2.36 [1.93 to 2.82]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; [analysis description as in outcome 1, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.70 to 1.27] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

3. Primary Outcome: Incidence Rate of Stroke or Systemic Embolism
Description: Incidence rate of stroke or systemic embolism on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.69 [0.45 to 0.94] | 1.01 [0.76 to 1.30]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; [analysis description as in outcome 1, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.43 to 1.06] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

4. Primary Outcome: Incidence Rate of Stroke
Description: Incidence rate of stroke on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only. Stroke is an acute onset of a focal neurological deficit of presumed vascular origin lasting for 24 hours or more or resulting in death. The stroke included ischemic or hemorrhagic or uncertain classification.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.64 [0.42 to 0.89] | 0.96 [0.70 to 1.22]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; [analysis description as in outcome 1, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.43 to 1.09] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

5. Primary Outcome: Incidence Rate of Transient Ischaemic Attack (TIA)
Description: Incidence rate of transient ischaemic attack (TIA) on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.30 [0.16 to 0.47] | 0.26 [0.12 to 0.41]

6. Primary Outcome: Incidence Rate of Systemic Embolism (SEE)
Description: Incidence rate of systemic embolism (SEE) on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.07 [0.00 to 0.16] | 0.06 [0.00 to 0.14]

7. Primary Outcome: Incidence Rate of Pulmonary Embolism (PE)
Description: Incidence rate of pulmonary embolism (PE) on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.09 [0.02 to 0.18] | 0.06 [0.00 to 0.14]

8. Primary Outcome: Incidence Rate of Major Bleeding Events
Description: Incidence rate of major bleeding events on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only. Major bleeding was defined as meeting one or more of the following criteria: Overt bleeding associated with a reduction in haemoglobin of at least 20 grams per liter or leading to a transfusion of at least 2 units of blood or packed cells; Symptomatic bleeding in a critical area or organ: Intraocular, intracranial, intraspinal or intramuscular with compartment syndrome, retroperitoneal bleeding, intra-articular bleeding or pericardial bleeding; Life-threatening bleeding.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.73 [0.49 to 0.98] | 1.42 [1.09 to 1.75]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous myocardial infarction, abnormal kidney function, concomitant antiplatelets use and concomitant use of drugs related to bleeding; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.38 to 0.88] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

9. Primary Outcome: Incidence Rate of Life-threatening Bleeding Events
Description: Incidence rate of life-threatening bleeding events on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only. Life-threatening bleeding was defined as meeting one or more of the following criteria: Symptomatic intracranial bleed; Reduction in haemoglobin of at least 50 grams per liter; Transfusion of at least 4 units of blood or packed cells, associated with hypotension requiring the use of intravenous inotropic agents; Necessitated surgical intervention; Fatal bleeding.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.50 [0.31 to 0.71] | 1.04 [0.77 to 1.34]

10. Primary Outcome: Incidence Rate of Vascular Death
Description: Incidence rate of vascular death on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.76 [0.51 to 1.02] | 1.00 [0.73 to 1.29]

11. Primary Outcome: Incidence Rate of Myocardial Infarction
Description: Incidence rate of myocardial infarction on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 0.34 [0.18 to 0.53] | 0.45 [0.27 to 0.64]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; A multivariable Cox regression model was performed including variables of treatment, age, gender, prior bleed, previous myocardial infarction, concomitant antiplatelets use, concomitant use of drugs related to bleeding, hypertension, and diabetes; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.49 to 1.84] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

12. Primary Outcome: Incidence Rate of All-cause Death
Description: Incidence rate of all-cause death on restricted set that included Dabigatran etexilate (DE) and Vitamin K Antagonist (VKA) only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Dabigatran Etexilate - Baseline | Vitamin K Antagonist (VKA) - Baseline
Number analyzed (Participants) | 1946 | 2509
Events per 100 person-years | 2.08 [1.69 to 2.51] | 3.27 [2.80 to 3.77]
Statistical Analysis 1: Comparison: Dabigatran Etexilate - Baseline vs Vitamin K Antagonist (VKA) - Baseline; [analysis description as in outcome 1, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.60 to 1.01] — Hazard ratio of dabigatran versus vitamin K antagonist (vitamin K antagonist as reference)

ADVERSE EVENTS:
Time Frame: From baseline visit until study completion or discontinuation, up to 3 years of follow-up.
Description: Enrolled and treated: All patients entered in the electronic data capture system who signed the informed consent and treated with at least once with the study treatments. Patients who were prescribed the combinations of oral anticoagulants at enrollment were excluded as no specific treatment can be defined for this group. For patients from the 'No treatment-initial' group, only their adverse events that happened when receiving certain treatment were reported in the respective treatment group.
Groups:
- Dabigatran Etexilate - at Least Once During the Study: All patients received at least once dabigatran etexilate during the study were included in the group. Adverse events which happened when the patients received dabigatran etexilate were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Vitamin K Antagonist (VKA) - at Least Once During the Study: All patients received at least once Vitamin K Antagonist (VKA) during the study were included in the group. Adverse events which happened when the patients received Vitamin K Antagonist (VKA) were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Rivaroxaban - at Least Once During the Study: All patients received at least once Rivaroxaban during the study were included in the group. Adverse events which happened when the patients received Rivaroxaban were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Apixaban - at Least Once During the Study: All patients received at least once Apixaban during the study were included in the group. Adverse events which happened when the patients received Apixaban were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Edoxaban - at Least Once During the Study: All patients received at least once Edoxaban during the study were included in the group. Adverse events which happened when the patients received Edoxaban were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse event happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Acetylsalicylic Acid (ASA) - at Least Once During the Study: All patients received at least once Acetylsalicylic acid (ASA) during the study were included in the group. Adverse events which happened when the patients received Acetylsalicylic acid (ASA) were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
- Antiplts Other Than ASA - at Least Once During the Study: All patients received at least once Antiplts other than Acetylsalicylic acid (ASA) during the study were included in the group. Adverse events which happened when the patients received Antiplts other than ASA were reported in this group.
  Patients can take any Antithrombotic treatments during the study. Adverse events were reported in the treatment group a patient actually received when the adverse events happened. Hence, the treatment groups in the adverse events section are not mutually exclusive.
Arm/Group | Dabigatran Etexilate - at Least Once During the Study | Vitamin K Antagonist (VKA) - at Least Once During the Study | Rivaroxaban - at Least Once During the Study | Apixaban - at Least Once During the Study | Edoxaban - at Least Once During the Study | Acetylsalicylic Acid (ASA) - at Least Once During the Study | Antiplts Other Than ASA - at Least Once During the Study
All-Cause Mortality (participants affected / at risk) | 116/2385 | 264/3258 | 166/2576 | 207/2934 | 17/368 | 141/1940 | 33/427
Serious Adverse Events (participants affected / at risk) | 79/2385 | 157/3258 | 92/2576 | 99/2934 | 10/368 | 70/1940 | 14/427
Other Adverse Events (participants affected / at risk) | 0/2385 | 0/3258 | 0/2576 | 0/2934 | 0/368 | 0/1940 | 0/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate - at Least Once During the Study (N=2385) | Vitamin K Antagonist (VKA) - at Least Once During the Study (N=3258) | Rivaroxaban - at Least Once During the Study (N=2576) | Apixaban - at Least Once During the Study (N=2934) | Edoxaban - at Least Once During the Study (N=368) | Acetylsalicylic Acid (ASA) - at Least Once During the Study (N=1940) | Antiplts Other Than ASA - at Least Once During the Study (N=427)
Anaemia (Blood and lymphatic system disorders) | 4 | 7 | 7 | 11 | 1 | 6 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 0 | 0 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 4 | 0 | 2 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2 | 1 | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Discoloured vomit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 10 | 14 | 6 | 2 | 12 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 6 | 4 | 1 | 1 | 3 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 2 | 4 | 1 | 1 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 12 | 7 | 5 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting projectile (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2
Medical device site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 2 | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 0 | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 5 | 0 | 0 | 0 | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 5 | 1 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Occult blood (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 8 | 2 | 3 | 1 | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 4 | 2 | 1 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 3 | 4 | 3 | 0 | 0 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 7 | 5 | 3 | 4 | 0 | 3 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 6 | 3 | 4 | 0 | 3 | 0
Vascular dementia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 8 | 6 | 5 | 0 | 2 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 4 | 1 | 0 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 16 | 6 | 7 | 1 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 8 | 1 | 4 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 4 | 1 | 3 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Subgaleal haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The data used in this analysis included only patients participating in Phase III of this study. Patients participating in Phase II were reported and analyzed in the 1160.129 phase II report, and were not planned to be reported separately for 1160.136.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01671007/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT01671007/SAP_001.pdf